CLINICAL TRIAL: NCT01731223
Title: Group Treatment for Insomnia in Primary Health Care: a Randomized Controlled Trial
Brief Title: Group Treatment for Insomnia in Primary Health Care
Acronym: Sleep Prime
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeanette Westman (Other)
Collaborators: Region Stockholm (Other Government); Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Jeanette Westman, PhD, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CeFAM, Karolinska Institutet
Record Dates: First submitted 2012-11-16; First posted 2012-11-21 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Insomnia
Keywords: Insomnia; Primary health care
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group treatment for insomnia (Experimental): Group treatment for insomnia.
  Interventions: Behavioral: Group treatment for insomnia
- No intervention (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Group treatment for insomnia — Experimental: Group treatment of insomnia The intervention is a group treatment based on cognitive and behavioral changing methods. It is including seven sessions during 10 weeks. Each session last for 2 hours with a 20 minutes pause. The intervention includes psycho education about sleep. Methods as relaxation, coping with worry, sleep restriction, stimulus control, sleep hygiene, stress coping strategies, strategies for coping with daytime symptom, identify and reformulate negative and dysfunctional thoughts about sleep, daytime functioning and stress and strategies for reducing hypnotics.
  Arms: Group treatment for insomnia

SUMMARY:
The aim of this study is to analyze if group treatment is effective to treat insomnia in primary healthcare.

DETAILED DESCRIPTION:
Insomnia is a common health problem. Untreated insomnia may lead to decreased physical and mental health. The patients turns to Primary Health Care when daytime symptoms decrease social and occupational function. Previous studies have shown that cognitive and behavioral therapy have effects on insomnia and recommends as first line treatment but is not widely available in primary health care.

The purpose is to test the effect of group intervention in Primary Health Care for patients with insomnia. The outcomes is insomnia severity, sleep habits, use of hypnotics, Fatigue, general health and health related quality of life. Characters with insomnia visiting in Primary Health Care.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia symptoms regarding DSM-V
* Motivated to group treatment.

Exclusion Criteria:

* Insomnia Severity Index less than 7 points
* Presence of acute life crises, acute psychiatric illness, bipolar disorder
* Shift work
* Linguistic or cognitive difficulties causing inability participate in group or fill in forms
* Insomnia directly caused by medical illness. Other sleep disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2010-08; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Insomnia severity Index | One year
  Insomnia Severity Index (ISI)is a seven item self assessment scale measuring severity of insomnia symptoms during the last two weeks. The items asks about sleep disturbance, daytime functioning and worrying about sleep. The possibly response is 0 "None" 1 "Mild" 2 "Moderate" 3 "Severe" 4 "Very severe". The sum is added and 0-7 p grades the insomnia to "none clinically significant insomnia", 8-14 p "subtreshold insomnia", 15-21 p "moderate insomnia", 22-28 p "severe insomnia".

SECONDARY OUTCOMES:
Fatigue severity scale | one year
  Measures fatigue symptoms in a seven item self assessment scale. Response from 1-7 points

OTHER OUTCOMES:
Sleep Logg | one year
  Sleep log for every night during two weeks. The patient logs time going to bed, sleep latency, awakes during the night, time going up from bed in the morning, total sleep time, sleep quality graded from 1-5. ! is very bad and 5 is very good). Use of alcohol, hypnotics and herbs are noted

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Westman, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Centre for family medicine, Stockholm, Huddinge
  - Centrum för allmanmedicin, Stockholm, Huddinge

REFERENCES:
- [Background] LeBlanc M, Beaulieu-Bonneau S, Merette C, Savard J, Ivers H, Morin CM. Psychological and health-related quality of life factors associated with insomnia in a population-based sample. J Psychosom Res. 2007 Aug;63(2):157-66. doi: 10.1016/j.jpsychores.2007.03.004. PMID 17662752
- [Background] Wilson SJ, Nutt DJ, Alford C, Argyropoulos SV, Baldwin DS, Bateson AN, Britton TC, Crowe C, Dijk DJ, Espie CA, Gringras P, Hajak G, Idzikowski C, Krystal AD, Nash JR, Selsick H, Sharpley AL, Wade AG. British Association for Psychopharmacology consensus statement on evidence-based treatment of insomnia, parasomnias and circadian rhythm disorders. J Psychopharmacol. 2010 Nov;24(11):1577-601. doi: 10.1177/0269881110379307. Epub 2010 Sep 2. PMID 20813762
- See also: Related Info — http://www.cefam.se